CLINICAL TRIAL: NCT02517905
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Local Administration of EXPAREL for Prolonged Postsurgical Analgesia in Subjects Undergoing Third Molar Extraction
Brief Title: Evaluation of EXPAREL for Prolonged Postsurgical Analgesia in Subjects Undergoing Third Molar Extraction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Collaborators: Lotus Clinical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 402-C-329
Record Dates: First submitted 2015-07-19; First posted 2015-08-07 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Dental Pain
MeSH Terms: conditions — Toothache | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EXPAREL 133 mg (Experimental): 10 mL EXPAREL (bupivacaine liposome injectable suspension) injected into the maxilla (4 mL; 2 mL per side) and mandible (6 mL; 3 mL per side) at the end of surgery and ≥20 min after lidocaine administration
  Interventions: Drug: Bupivacaine liposome
- Placebo (Placebo Comparator): 10 mL normal saline injected into the maxilla (4 mL; 2 mL per side) and mandible (6 mL; 3 mL per side) at the end of surgery and ≥20 min after lidocaine administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacaine liposome — Local administration
  Other Names: EXPAREL
  Arms: EXPAREL 133 mg
Drug: Placebo — Local administration
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, double-blind, placebo-controlled study in subjects scheduled to undergo elective bilateral third molar extraction under local anesthesia. At least one lower mandibular third molar must involve full or partial bony impaction confirmed by visual or radiographic evidence.

DETAILED DESCRIPTION:
Subjects will be screened within 30 days prior to surgery.

Randomized subjects will receive a dental nerve block with lidocaine 2% with epinephrine 1:100,000 before undergoing bilateral third molar extraction under local anesthesia. In addition to the lidocaine nerve block, the Investigator may choose to add topical benzocaine or intraoperative nitrous oxide.

At the end of surgery, and at least 20 minutes after the lidocaine administration, blinded study drug will be infiltrated to provide postsurgical analgesia. Subjects will be required to remain in the research facility for 96 hours after study drug administration.

Postsurgical efficacy, safety, and pharmacokinetic (PK) assessments will be conducted.

All subjects will return for a follow-up visits on Days 7 and 10. A phone call will be made to each subject on Day 30 for an adverse event (AE) assessment and to inquire as to whether the subject made any unscheduled phone calls or office visits related to pain.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years of age at screening.
2. Scheduled to undergo bilateral third molar extractions (i.e., extraction of all four third molars) under local anesthesia. At least one lower mandibular third molar must involve full or partial bony impaction confirmed by visual or radiological evidence.
3. American Society of Anesthesiology (ASA) physical status 1, 2, or 3.
4. Female subjects must be either surgically sterile, using a medically acceptable method of birth control, or at least 2 years postmenopausal, and must have a documented negative pregnancy test result during screening and on Day 1 prior to surgery.
5. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics or opioids.
2. Contraindication to lidocaine, epinephrine, bupivacaine, or oxycodone.
3. History of significant drug allergy (e.g., anaphylaxis or hepatotoxicity).
4. Positive test result from the urine drug screen at screening or prior to the surgical procedure.
5. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration.
6. History or active psychiatric illness (including major depression, bipolar disorder, or anxiety); Type 1 or Type 2 diabetes; severe renal or hepatic impairment; significant cardiovascular disease (including cardiac rhythm disturbance); migraine headaches, frequent headaches, other pain conditions, or other medical condition that, in the opinion of the Investigator, may increase the risk of surgery or interfere with the evaluation of the study drug.
7. History of infection requiring intravenous (IV) antibiotics within 45 days or oral (PO) antibiotics within 30 days prior to study drug administration for reasons other than dental prophylaxis. Subjects must be afebrile, without signs or symptoms indicative of active infection.
8. Use of any of the following medications within the times specified before surgery: long-acting opioid medication, nonsteroidal anti-inflammatory drugs (NSAIDs), aspirin (except for low-dose aspirin used for cardioprotection), or acetaminophen within 3 days, or any opioid medication within 24 hours.
9. Initiation of treatment with any of the following medications within 1 month of EXPAREL infiltration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®). If a subject is taking one of these medications for a reason other than pain control, he or she must be on a stable dose for at least 1 month prior to EXPAREL administration.
10. Current use of systemic glucocorticosteroids within 1 month of enrollment in this study.
11. Use of any concurrent therapy that could interfere with the evaluation of efficacy or safety, such as any drugs which in the Investigator's opinion may exert significant analgesic properties or act synergistically with the investigational product.
12. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Jones, MD, PharmD, Study Director — Pacira Pharmaceuticals, Inc
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EXPAREL 133 mg | Placebo
Started | 107 | 59
Completed | 97 | 57
Not Completed | 10 | 2
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Screen failure | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received study drug, with analysis by actual treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | EXPAREL 133 mg | Placebo | Total
Number analyzed (Participants) | 105 | 57 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.9 (3.81) | 20.9 (4.76) | 20.9 (4.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 33 | 86
  Male | 52 | 24 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 7 | 23
  Not Hispanic or Latino | 89 | 50 | 139
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 1 | 10
  White | 94 | 53 | 147
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 105 | 57 | 162
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.8 (6.87) | 24.5 (4.72) | 25.3 (6.21)
Impaction Scores [Count of Participants; unit: Participants]
  4 fully bony impacted teeth | 23 | 19 | 42
  3 fully bony impacted teeth, 1 partially impacted | 14 | 7 | 21
  3 fully bony impacted teeth | 1 | 3 | 4
  2 fully bony impacted teeth, 2 partially impacted | 10 | 7 | 17
  2 fully bony impacted teeth, 1 partially impacted | 9 | 2 | 11
  2 fully bony impacted teeth | 3 | 6 | 9
  1 fully bony impacted tooth, 3 partially impacted | 4 | 1 | 5
  1 fully bony impacted tooth, 2 partially impacted | 7 | 3 | 10
  1 fully bony impacted tooth, 1 partially impacted | 8 | 5 | 13
  1 fully bony impacted tooth | 2 | 2 | 4
  4 partially impacted teeth | 3 | 0 | 3
  3 partially impacted teeth | 4 | 0 | 4
  2 partially impacted teeth | 16 | 1 | 17
  1 partially impacted tooth | 1 | 1 | 2
  No impactions | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Numeric Rating Scale (NRS) Pain Intensity Scores Through 48 Hours
Description: AUC of NRS pain intensity scores through 48 hours. Pain intensity scores were measured on a 10-point scale (0=no pain and 10=worst possible pain)
Time Frame: 0-48 hours
Population: Primary efficacy population: all participants who received study drug, underwent the surgery, and were enrolled under protocol amendment 2, according to which pain intensity scores were collected before each use of rescue medication. Analysis was based on randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: units on NRS scale*hr
Arm/Group | EXPAREL 133 mg | Placebo
Number analyzed (Participants) | 99 | 51
units on NRS scale*hr | 178.9 (10.30) | 181.6 (13.63)
Statistical Analysis 1: Comparison: EXPAREL 133 mg vs Placebo; Test type: Superiority; p = 0.8661, ANOVA; LSMD = -2.7, 95% CI 2-sided [-33.5 to 28.2]

2. Secondary Outcome: Area Under the Curve (AUC) of Numeric Rating Scale (NRS) Pain Intensity Scores Through 24 Hours
Description: AUC of NRS pain intensity scores through 24 hours. Pain intensity scores were measured on a 10-point scale (0=no pain and 10=worst possible pain) 0-24 hours
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on NRS scale*hr
Arm/Group | EXPAREL 133 mg | Placebo
Number analyzed (Participants) | 99 | 51
units on NRS scale*hr | 102.4 (4.73) | 106.4 (6.26)
Statistical Analysis 1: Comparison: EXPAREL 133 mg vs Placebo; Test type: Superiority; p = 0.5780, ANOVA; LSMD = -4.0, 95% CI 2-sided [-18.2 to 10.2]

3. Secondary Outcome: Area Under the Curve (AUC) of Numeric Rating Scale (NRS) Pain Intensity Scores Through 72 Hours
Description: AUC of NRS pain intensity scores through 72 hours. Pain intensity scores were measured on a 10-point scale (0=no pain and 10=worst possible pain)
Time Frame: 0-72 hours
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: units on NRS scale*hr
Arm/Group | EXPAREL 133 mg | Placebo
Number analyzed (Participants) | 99 | 51
units on NRS scale*hr | 241.5 (15.40) | 235.6 (20.38)
Statistical Analysis 1: Comparison: EXPAREL 133 mg vs Placebo; Test type: Superiority; p = 0.8010, ANOVA; LSMD = 5.9, 95% CI 2-sided [-40.2 to 52.1]

4. Secondary Outcome: Percentage of Opioid-free Subjects Through 24 Hours.
Description: Percentage of opioid-free subjects through 24 hours.
Time Frame: 0-24 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EXPAREL 133 mg | Placebo
Number analyzed (Participants) | 99 | 51
Participants | 19 | 12

5. Secondary Outcome: Percentage of Opioid-free Subjects Through 48 Hours.
Description: Percentage of opioid-free subjects through 48 hours.
Time Frame: 0-48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EXPAREL 133 mg | Placebo
Number analyzed (Participants) | 99 | 51
Participants | 19 | 12

6. Secondary Outcome: Percentage of Opioid-free Subjects Through 72 Hours.
Description: Percentage of opioid-free subjects through 72 hours.
Time Frame: 0-72 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EXPAREL 133 mg | Placebo
Number analyzed (Participants) | 99 | 51
Participants | 18 | 12

ADVERSE EVENTS:
Time Frame: From screening to postsurgical day 29
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (eg abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug without any judgment about causality. Serious AEs were defined as per clinicaltrials.gov.
  The safety analysis set included all subjects who received study drug, based on the treatment received.
Arm/Group | EXPAREL 133 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/57
Other Adverse Events (participants affected / at risk) | 105/105 | 57/57
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL 133 mg (N=105) | Placebo (N=57)
Hypoesthesia oral (Nervous system disorders) | 104 | 57
Dysgeusia (Nervous system disorders) | 80 | 32
Muscle contractions involuntary (Nervous system disorders) | 16 | 12
Dizziness (Nervous system disorders) | 11 | 8
Headache (Nervous system disorders) | 6 | 9
Paresthesia oral (Nervous system disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 32 | 16
Vomiting (Gastrointestinal disorders) | 18 | 9
Alveolar osteitis (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Post procedural edema (Injury, poisoning and procedural complications) | 10 | 7
Post procedural swelling (Injury, poisoning and procedural complications) | 3 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 8 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Wound infection (Infections and infestations) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hot flush (General disorders) | 1 | 2
Blurred Vision (Eye disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site shall reasonably cooperate with the sponsor to prepare an abstract and/or manuscript reporting trial results within 90 and 120 days, respectively, after final CSR is available and should not otherwise publish any results within 120 days. Scientific meeting and journal are to be determined by the sponsor. Site shall give sponsor ≥60 days before submitting materials and upon sponsor request shall withhold publication for an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2015-09-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT02517905/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT02517905/SAP_001.pdf